CLINICAL TRIAL: NCT06428305
Title: The Effect of Hygiene Education Given Using the Teach-Back Method to Pregnant Women Diagnosed With Urinary Tract Infections on Hygiene Behaviors and Symptoms: A Randomized Controlled Trial
Brief Title: Providing Hygiene Education Using the Teach-back Method to Pregnant Women Diagnosed With Urinary Tract Infections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Responsible Party: Principal Investigator, Arzu Çiftçi, Graduate student, KTO Karatay University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: KARATAYU-EBE-AÇ-01
Record Dates: First submitted 2024-05-20; First posted 2024-05-24 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Urinary Tract Infections During Pregnancy
Keywords: Pregnant; Genital hygiene; Teach Back Method; Health Educatio; Urinary system ınfections

STUDY DESIGN:
Intervention Model Description: The intervention group receiving planned education on genital hygiene using the teach-back method and the control group not receiving education
Who Masked: Participant, Outcomes Assessor
Masking Description: The statistician will be blinded in the research. Researcher blinding cannot be done because he is a practitioner. But the researcher will open the envelope created by the statistician just before the application and find out which group the mother belongs to. In order to prevent bias in the evaluation of the data, groups will be coded as A and B, and the analysis of the data will be carried out by an independent statistical expert. After the analysis and interpretation of the data are completed, the codes of the intervention and control groups of the study will be revealed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The intervention group receiving planned education on genital hygiene using the teach-back method (Experimental): All pregnant women diagnosed with UTI at the maternity outpatient clinic are prescribed antibiotics containing the active substance fosfomycin tromethamol, which is recommended for uncomplicated urinary tract infections of adults. The duration of the antibiotic's effect is seven days (Due date). After completing the treatment process determined according to the physician's request, training and counseling will be provided using the Genital Hygiene Training Guide based on the Tell me what you have learned method. In this context, 4 interviews will be held during the project.
  Interventions: Other: Providing hygiene education based on the method of teaching what has been learned in the context of a genital hygiene guide
- Control Group (No Intervention): Control Group: Research data were collected from pregnant women who were in the control group at the December intervals with the experimental group, as shown in the Flow Chart of the study. After the completion of the study, this group will also be given an education and training booklet.

INTERVENTIONS:
Other: Providing hygiene education based on the method of teaching what has been learned in the context of a genital hygiene guide — As shown in the Flow Chart of the study, research data were collected from pregnant women who were in the control group at the December intervals with the experimental group. After the completion of the study, this group will also be given an education and training booklet.
  Arms: The intervention group receiving planned education on genital hygiene using the teach-back method

SUMMARY:
This study proves that the hygiene education given to pregnant women diagnosed with tract infection by explaining what they have learned increases the duration of genital health, thus ensuring the positive health development of women and protecting and improving their health. At the same time, it is aimed to inform the professional "tell what you have learned" method and to guide the practices of those working in the field of health. The research will be conducted in a randomized control design with a pretest-posttest control group. The population of the research will consist of pregnant women who were followed up in the relevant hospital and who met the inclusion criteria on the dates the research was conducted. The number of samples for the study was determined as 36 participants, 18 in each group. While hygiene training will be given to the intervention group using the tell-what-you-learned method, no training will be given to the control group. Personal Information Form and Genital Hygiene Behavior Scale will be used as data collection tools in the research. Data will be collected at the first encounter, day 7, day 21, and day 30. In evaluating the data, the suitability of the variables to normal distribution will be examined using visual analytical methods. When comparing application results within and between groups, parametric or nonparametric tests will be used depending on whether they show a normal distribution or not, and t test or Mann-Withney U Test will be used to compare the difference between two groups. Wilcoxon test will be used to analyze pre- and post-intervention results within the same group. Statistical significance level will be accepted as p<0.05. When the literature is examined, there are studies on different health education plans for women diagnosed with urinary tract infection during pregnancy, but since there is no research on the tell-what-you-learned method, it is an original study, and at the same time, the previous knowledge levels of pregnant women diagnosed with UTI were learned and the effect of the education given on their behavior was examined. It is thought that this teaching method will contribute positively to the knowledge level and behavior of women.

DETAILED DESCRIPTION:
Urinary tract infection in women is the second most common discomfort after anemia that occurs during certain periods of life during pregnancy and is also one of the most common bacterial infections (Fihn, 2003; Griebling, 2005; Czajkawski, Bras-Konopeielka and Teliga-Czajkowska, 2021). About 50% of women have urinary tract infections at least once in their lifetime (Gilbert, O'bien, Hutgen et al., 2013). In the presence of urinary tract infection, painful urination is usually observed, frequent emergency toilet trips, while other symptoms include lower abdominal or pelvic pain and pressure, blood in the urine, milky, cloudy or pink/red urine color, fever, heavily scented urine, nausea, vomiting and diarrhea (Habak and Griggs Dec, 2023). Pregnancy, number of pregnancies, age, diabetes mellitus, urethrogenital anomalies, genetic and behavioral factors, hygiene deficiency, anemia, history of urinary system infection (Bekzac, Orgul, Tanacan et al., 2019), factors such as low socio-economic level, inadequate perineal hygiene, vaginal douching, long-term use of antibiotics and steroids, smoking, alcohol consumption and immune deficiencies increase the incidence (Özdemir, Ortabağ, Tosun et al., 2012; Ejder Apay, Özdemir, Nazik et al., 2014; Karahan, 2017). The frequency of sexual experience, the number of sexual partners (current or previous years), not urinating after sexual intercourse, the direction of wiping the perineum after the toilet, urine retention, daily insufficient water consumption also play an important role (Seid, Markas, Aklilu et al., 2023).

Physiological, anatomical and hormonal changes experienced during pregnancy increase the predisposition to urinary tract infection (Helli, Dolapçıoğlu and Hammer, 2011). Urinary tract infection has a prevalence rate of 20% among pregnant women (Abdel- Deciz Elzayat, Barnett-Vanes, Dabour et al., 2013; Salari, Khoshbakht, Hemmati et al., 2023). Approximately 5-12% of pregnant women are affected by asymptomatic bacteria, while 30% of women with symptoms may develop cystitis or 50% pyelonephritis. Asymptomatic bacteriuria can lead to many undesirable maternal and neonatal problems if left untreated (De Oliveira Neto et al., 2021). Preeclampsia can cause undesirable consequences such as hypertensive diseases, pyelonephritis, permanent kidney damage, anemia, premature rupture of membranes, premature birth threat, low birth weight, fetal deaths and cesarean section (Lawani, Alade and Oyelaran, 2015; Willy, Wanyoike and Mugo, 2015). These are conditions that cause many physiological and anatomical damages and are common, requiring urgent treatment (Sevil, Özdemir, Aleattin et al., 2013; Apay, Özdemir, Nazik et al., 2014; Karahan, 2017). In addition, more than half of the patients complain of clinical depression and 38.5% of them complain of anxiety. It is reported that significant improvement in quality of life has been observed after appropriate treatment and prophylaxis (Renard, Ballarini, Mascarenhas et al., 2015). It is an important public health problem and can negatively affect the life of women and families, causing deterioration of the quality of life (Sevil, Özdemir, Aleattin et al., 2013; Apay, Özdemir, Nazik et al., 2014; Karahan, 2017). It causes a significant financial impact of up to billions of dollars on both the health system and society (Akram, Shahid and Khan, 2007; Martini, Horner, Roehrs et al., 2007; De Oliveira Neto et al., 2021). Therefore, it is important to plan and implement initiatives aimed at improving and preventing urinary tract infections.

When the studies were examined, it was found that incorrect, incomplete or faulty hygiene behaviors increased the incidence of urinary tract infections (Özdemir et al., 2012; Sevil et al., 2013; Karahan, 2017). In urinary tract infections, it is necessary to determine the wrong behaviors first about hygiene and to provide permanent and positive behavioral changes by providing trainings for them (Karahan, 2017).

Genital hygiene behaviors are an important factor in the formation and prevention of urinary tract infections. Öner and Çeber Turfan (2020) stated that in addition to medical treatment, urinary tract infection symptoms can be prevented with hygiene education and that it also positively affects genital hygiene behaviors (Öner and Çe October Turfan, 2020). Regarding the educational methods, Sinan et al. A study conducted by (2020) concluded that genital infection awareness training based on the knowledge-motivation-behavior skills model increases women's knowledge level and positively reinforces women's hygiene behaviors (Sinan, Kaplan, Sahin et al., 2020). In another study conducted on genital hygiene behavior training given using audiovisual and brochure, it was found that the intervention group developed more positive behaviors than the control group (Hayati et al., 2018). Parlas and Eryilmaz (2023) It is stated that the knowledge, attitudes and behaviors of women who receive education based on the PRECEDE-PROCEED model are positively affected (Parlas & Eryilmaz, 2023). In particular, in another study, it is stated that planned education and home visits on genital hygiene have a positive effect (Abic, Yatmaz, Altınışık et al., 2024). In addition, web-based genital hygiene education has a positive effect on self-care power and genital hygiene behaviors (Gül and Yağmur, 2023), peer education provided under the guidance of the health improvement model is effective and increases the knowledge levels of young October adults about genital hygiene behaviors (Polat, Küçükkelepçe et al., 2022) is stated. Another study conducted to determine the effect of genital hygiene education given by three different methods, oral education after medical curettage, education with written material and just demonstration on genital hygiene behaviors, found that oral education alone is not effective in providing and developing genital hygiene behaviors, and the demonstration method is more effective than oral and written education methods (Uzun and Göktaş, 2022). As a result of the current literature review, although the importance of genital hygiene education is emphasized, it is clear that there is a need for teaching techniques that will provide permanent behavioral changes. Midwives, who are in contact the most during the pregnancy period and conduct face-to-face interviews, undertake the most important task in teaching genital hygiene behaviors effectively and correctly (Ünsal, Özyazıcıoğu, Sezgin et al. 2010). For this reason, midwives should plan training with a permanent teaching technique that fills in gaps in the lack of knowledge, can get feedback, can be evaluated, while advising pregnant women diagnosed with urinary tract infection on genital hygiene behaviors.

The teach back method is a method used for the education, learning, evaluation and development of personal care behaviors of individuals. This approach provides an opportunity for individuals to understand educational materials, improve their level of retention in mind, and evaluate themselves. One of the important advantages is that the educational content is presented as simply as possible, free from medical terms, and that the clients repeat the practices at the end of the training (Ahmed Abd El- hamed, 2023). The practice involves asking patients by a health professional to explain in their own sentences what they have just been told. If there is any misunderstanding, it is clarified by the health professional and the understanding status is evaluated by checking again. This condition continues until the patient tells the truth and remembers the information given to him (Farris, 2015; Talevski, Wong Shee, Rasmussen et al., 2020). The patient's learning about issues related to health information can be improved through continuous feedback. It is stated that this method-based communication approach helps patients to better understand their own medical conditions and health information, and provides benefits in improving their skills of remembering and applying medical information (Tamura, 2013; Laws, 2018; Cheng, Chen, 2023).The Tell what you have learned method provides positive effects on information acquisition, remembering, keeping in mind, as well as health behavior management, personal care behavior development, hospitalization, quality of life and patient satisfaction (Yen and Leasure, 2019; Talevski et al., 2020; Cheng et al., 2023). In addition, it is stated that self-care increases strength and comfort, reduces the cost of health care (Badeczewski et al., 2017; Imanipour, Molazem, Rakhshan et al., 2022). For this reason, midwives can use the tell what you've learned method, which is a permanent teaching technique that fills in gaps in the lack of information, can be reversed, evaluated, while advising pregnant women diagnosed with urinary tract infection on genital hygiene behaviors.

Pregnant women diagnosed with urinary tract infection have been given trainings on genital hygiene behaviors in many different methods in the literature, but when the trainings given were examined, it was determined that teaching techniques aimed at improving the education, learning level, evaluation and personal care behaviors of individuals are needed. It is thought that using the tell what you have learned method in order to fill these gaps in education will be beneficial. In this context, the fact that there are no studies on the subject in our country, the fact that evidence-based teaching techniques are tried in new areas constitutes the original value of the project and our main motivation. The project has unique value for a sustainable future in terms of its effects on pregnant women in particular and qualified midwifery care at the social level in general. It will also enable data to be obtained for comparing innovative educational methods with traditional educational methods. Thus, it will help to improve, organize or develop capacity for future initiatives.

Hypotheses

1. The education given to pregnant women who have been diagnosed with urinary tract infection by the tell me what you have learned method positively affects genital hygiene behavior.
2. Education given to pregnant women who have been diagnosed with urinary tract infection by the tell-what-you-learned method reduces the level of symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Able to read and write Turkish,
* Those between the ages of 18-35 December,
* Diagnosed with urinary tract infection,
* Pregnant women who are open to communication (who are competent to understand and answer questions) will be included in the sample.

Exclusion Criteria:

* Leaving the research of his own accord,
* Having a diagnosis related to risky pregnancy other than the diagnosis of urinary tract infection
* With a history of psychiatric illness (self-report),
* Pregnant women with a history of gynecological diseases (self-information) will be excluded from the research.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant women who have been diagnosed with a urinary tract infection
Enrollment: 36 (Actual)
Dates: Start 2024-04-22 (Actual); Primary Completion 2024-05-21 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
The Scale of Genital Hygiene Behaviors | 1. day, 7. day, 21, day, 30.. day
  It was developed by Karahan (2017) to evaluate genital hygiene behaviors in women. General hygiene habits (top 12 items), menstrual hygiene (13th item on the five-point likert scale).-20. substances) and abnormal finding awareness (21-23. it consists of three sub-dimensions (substances) and a total of 23 substances. The cronbach alpha value of the entire scale is 0.80, and it is stated that the general hygiene sub-dimension is 0.70, the menstrual hygiene sub-dimension is 0.74, and the abnormal finding awareness sub-dimension is 0.81. 7 of the scale., 14., 19., 20., 23. items are scored in reverse. The lowest 23 highest 115 points are taken from the scale and the high scores indicate that genital hygiene behavior is positive (Karahan, 2017).

CONTACTS AND LOCATIONS:
Overall Officials: Hediye KARAKOÇ, assistant professor, Study Director — KTO Karatay University; Arzu ÇİFTÇİ, post graduate, Principal Investigator — KTO Karatay University
Locations (1):
- KTO Karatay University, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
have no plans to make individual participant data (IPD) available to other researchers.